CLINICAL TRIAL: NCT04888013
Title: The Impact of Birth Environment and Childbirth-stress, Birth Control & Outcome
Brief Title: Birth Environment and Childbirth-stress, Control & Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Taoyuan General Hospital (Other Government)
Responsible Party: Principal Investigator, Li-li Chen, RN PhD student, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: TYGH109064
Record Dates: First submitted 2021-05-02; First posted 2021-05-17 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Childbirth Problems; Birth; Delayed
Keywords: birth Environment; childbirth-stress; birth control; outcomes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): Routine care for childbirth
  Interventions: Other: Positive Birth Environment
- experimental 2 (Experimental): Building childbirth environment
  Interventions: Other: Positive Birth Environment
- experimental 1 (Experimental): Building childbirth environment and labor delivery recovery room
  Interventions: Other: Positive Birth Environment

INTERVENTIONS:
Other: Positive Birth Environment — The intent is to surround the woman and her caregivers with specific types of auditory, visual, and tactile stim uli. One key feature of the ambient room is what is missing-the standard hospital bed. As an alternative, a portable double-sized mattress with several large pillows is set up in a corner of the room. The intent is to allow the woman freedom in positioning and to permit close contact with support people, and to limit the routine use of continuous elec tronic fetal heart rate monitoring and other technologies during normal labor. Lighting is dimmed. A wide variety of music selections are also available.

SUMMARY:
This research improves the correlation between birth control and birth outcomes by understanding the childbirth environment and birth stress. A Quasi Experiment research . The sample size was calculated using a two-tailed test, the significance level α was 0.05, the power was 80%, three groups of repeated measurements were taken three times, the effect size (effect size) was set to medium.25, and the required number of samples was 108 people, resulting in a 20% wastage rate, a total of 129 people are needed, so each of the three groups is expected to accept 43 people.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 20 years old,
2. Those who agree to participate in this research and can read and write Chinese,
3. vaginal delivery
4. Those who have no high-risk complications or chronic diseases during pregnancy and childbirth.

Exclusion Criteria:

1. Those who have been diagnosed with mental illness by a doctor, including those with depression and mood disorders
2. Exclude stillbirths and newborns with congenital abnormalities

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Stress Scale | From latent phase to postpartum 2 hours
  The visual analogue scale for stress is a horizontal line of 0-10 cm. It is divided into the maximum level of stress. 0 means no stress at all, and 10 means extreme stress. The individual will point out the most suitable value for the feeling at this moment. Centimeters represent one point, and fractions gradually represent a decrease in the score
salivary amylase | From latent phase to postpartum 2 hours
  he measurement standard values are as follows: 30 kIU/L is no pressure; 31~45 kIU/L is a small amount of pressure; 46~60 kIU/L is a moderate pressure; more than 61 kIU/L is a severe pressure.
Heart rate variability | From latent phase to postpartum 2 hours
  The heart rate variability measurement uses TS-0411 sample, wrist-type physiological monitor (approved by the Department of Health No. 5200277), with multiple built-in biological sensors, which have been calibrated before leaving the factory to achieve high accuracy.

SECONDARY OUTCOMES:
Perception of Childbirth Environment Scale | through study completion, an average of Postpartum 24 hours
  Using LIKERT-5, the higher the score, the better the environmental experience

CONTACTS AND LOCATIONS:
Overall Officials: Ll-li Chen, PhD Student, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Taoyuan General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ayerle GM, Schafers R, Mattern E, Striebich S, Haastert B, Vomhof M, Icks A, Ronniger Y, Seliger G. Effects of the birthing room environment on vaginal births and client-centred outcomes for women at term planning a vaginal birth: BE-UP, a multicentre randomised controlled trial. Trials. 2018 Nov 19;19(1):641. doi: 10.1186/s13063-018-2979-7. PMID 30454075
- [Result] Downe S, Finlayson K, Oladapo OT, Bonet M, Gulmezoglu AM. Correction: What matters to women during childbirth: A systematic qualitative review. PLoS One. 2018 May 17;13(5):e0197791. doi: 10.1371/journal.pone.0197791. eCollection 2018. PMID 29772012
- [Result] Hodnett ED, Stremler R, Weston JA, McKeever P. Re-conceptualizing the hospital labor room: the PLACE (pregnant and laboring in an ambient clinical environment) pilot trial. Birth. 2009 Jun;36(2):159-66. doi: 10.1111/j.1523-536X.2009.00311.x. PMID 19489810
- [Result] Lorentzen I, Andersen CS, Jensen HS, Fogsgaard A, Foureur M, Lauszus FF, Nohr EA. Study protocol for a randomised trial evaluating the effect of a "birth environment room" versus a standard labour room on birth outcomes and the birth experience. Contemp Clin Trials Commun. 2019 Feb 15;14:100336. doi: 10.1016/j.conctc.2019.100336. eCollection 2019 Jun. PMID 30886935